CLINICAL TRIAL: NCT02077569
Title: The Short Term Effects of an AKT Inhibitor (AZD5363) on Biomarkers of the AKT Pathway and Anti-tumour Activity in a Breast Cancer Paired Biopsy Study
Brief Title: AKT Inhibitor in Oestrogen Positive Breast Cancer
Acronym: STAKT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: AstraZeneca (Industry); Cancer Research UK (Other); National Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 12076
Record Dates: First submitted 2014-01-16; First posted 2014-03-04 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Invasive Breast Cancer
Keywords: AKT inhibitor; AZD5363; Anti-tumour activity; Breast cancer; ER positive; Oestrogen positive; post menopausal; chemotherapy required; no prior cancer treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — capivasertib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AZD5363 480mg (Experimental): STAGE 1 ONLY AZD5363 480mg Twice daily dosing for 4 and 1/2 days (9 doses) Oral Capsule
  Interventions: Drug: AZD5363
- Placebo (Placebo Comparator): STAGE 1 ONLY Twice daily dosing for 4 and 1/2 days (9 doses) Oral Capsule
  Interventions: Drug: AZD5363
- AZD360mg (Experimental): STAGE 2 AZD5363 360mg Twice daily dosing for 4 and 1/2 days (9 doses) Oral Capsule
  Interventions: Drug: AZD5363
- AZD5363 240mg (Experimental): STAGE 2 AZD5363 240mg Twice daily dosing for 4 and 1/2 days (9 doses) Oral Capsule
  Interventions: Drug: AZD5363

INTERVENTIONS:
Drug: AZD5363 — Stage 1: AZD5363 480mg or placebo twice daily oral dosing for 4 and 1/2 days (9 doses) Stage 2: AZD5363 360mg or 240mg daily oral dosing for 4 and 1/2 days (9 doses)

SUMMARY:
To compare the effect of four and a half days treatment of a range of doses of AZD5363 on selected markers of the AKT pathway and anti-proliferation compared with placebo in oestrogen receptor positive breast cancers.

To assess the tolerability of four and a half days treatment of AZD5363.

DETAILED DESCRIPTION:
The principal research questions to be addressed are whether (or not) AZD5363 is "hitting its therapeutic target" sufficiently and to the extent that is required to produce efficacy in pre-clinical experiments.

The primary endpoint markers have been selected to determine this.

Reductions in markers of the AKT pathway and increases in markers of anti-proliferation will characterise the degree of biological activity arising from the inhibition of AKT across a range of doses of AZD5363.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. WHO performance status 0-1.
3. Able to swallow & retain oral medication.
4. Patients who fall in to either category (a) or (b):

   1. Post-menopausal patients
   2. Pre-menopausal patients who also meet at least one of the criteria (i), (ii) or (iii) below:

   i) hysterectomy or bilateral fallopian tube ligation at least 6 weeks ago plus a negative pregnancy test.

   ii) true abstinence iii) willing to have pregnancy testing and use 2 forms of contraception
5. Female patients, aged 18 years and over, with histological confirmation of ER positive invasive breast carcinoma.
6. Stage 1/2/3 or Stage 4 with primary tumour in the breast amenable to biopsies. New primary breast tumours (ipsi- or contra-lateral) despite prior endocrine treatment for an earlier primary breast tumour with at least 12 months interval between cessation of endocrine therapy and Visit 1 are eligible.
7. Scheduled to have chemotherapy based on tumour characteristics and local treatment protocols.
8. Tumours large enough to provide sufficient tissue to be taken by core-cut or tru-cut biopsy to provide tissue sections for the marker assays.

Exclusion Criteria:

1. Prior treatment for breast cancer except new primary breast tumours arising despote prior endocrine treatment for an earlier primary breas tumour with at least 12 months interval between cessation of endocrine therapy and Visit 1 (see inclusion criteria 6).
2. Known ER negative tumour.
3. Female patients with histological confirmation of ER+ve invasive breast carcinoma not scheduled to have chemotherapy
4. Exposure to potent inhibitors or inducers of CYP3A4 or CYP2D6 or substrates of CYP3A4 within 2 weeks before the first dose of study treatment (3 weeks for St Johns Wort).
5. Clinically significant abnormalities of glucose metabolism
6. Major surgery (excluding placement of vascular access) within 4 weeks before the first dose of study treatment.
7. Spinal cord compression or brain metastases.
8. Evidence of severe or uncontrolled systemic disease.
9. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc)>450 msec obtained from 3 consecutive ECGs; - Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events.
   * Any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure NYHA Grade 2.
   * Uncontrolled hypotension.
10. Absolute neutrophil count <1.5 x 10,000,000,000/L
11. Platelet count <100 x 10,000,000,000/L.
12. Haemoglobin <90 g/L
13. ALT >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases.
14. Elevated ALP is not exclusionary if due to the presence of bone metastasis and liver function is otherwise considered adequate
15. Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of liver metastases.
16. Creatinine >1.5 times ULN concurrent with creatinine clearance <50 ml/min; confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN
17. Proteinuria >3+ on dipstick analysis.
18. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD5363.
19. History of hypersensitivity to active or inactive excipients of AZD5363 or drugs with a similar chemical structure or class to AZD5363.
20. Current disease or condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
21. Past medical history of interstitial lung disease, drug induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
22. Evidence of dementia, altered mental status or any psychiatric condition that would prohibit understanding or rendering of informed consent
23. Previous allogeneic bone marrow transplant.
24. Known immunodeficiency syndrome.
25. Pregnant or lactating patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: Pharmacodynamic biomarker analysis in tumour tissue to assess the biological effect of AZD5363 on markers of anti-proliferation and the AKT pathway | Up to 42 months: Stage 1: up to 60 participants in up to 20 months. Stage 1 biomarker analysis early in Stage 2. Stage 2 proceeds where reduction in 1 of the 3 primary biomarkers. Stage 2: up to 60 participants in up to 16 months.
  Changes in pPRAS40, pGSK3b, Ki67

SECONDARY OUTCOMES:
Compare anti-proliferative effect on markers of the AKT pathway after 4&1/2days treatment at 3 different doses of AZD5363 vs placebo in Er +ve breast cancers | Up to 42 months. Stage 1: up to 60 participants in up to 20 months. Stage 2: up to 60 participants in up to 16 months.
  By measuring biological changes in the tumour and circulation via measurement of changes in alternative biological markers which relate to the AKT pathway:
  Tumour total and pAKT Tumour: cleaved caspase 3; pS6 (IHC); FOXO3a Blood (platelet-rich plasma): Total and pPRAS40; Total and pGSK3b; Total and pAKT.
Compare direct effect on markers of the AKT pathway after 4&1/2days treatment at 3 different doses of AZD5363 vs placebo in Er +ve breast cancers | Up to 42 months. Stage 1: up to 60 participants in up to 20 months. Stage 2: up to 60 participants in up to 16 months.
  By measuring biological changes in the tumour and circulation via measurement of changes in alternative biological markers which relate to the AKT pathway:
  Tumour total and pAKT Tumour: cleaved caspase 3; pS6 (IHC); FOXO3a Blood (platelet-rich plasma): Total and pPRAS40; Total and pGSK3b; Total and pAKT.
To measure tolerability and toxicity following short term (four and a half days) exposure to AZD5363 | Up to 42 months. Stage 1: up to 60 participants in up to 20 months. Stage 2: up to 60 participants in up to 16 months.
  Tolerability and toxicity will be measured following short term exposure to AZD5363 by incidence and severity of adverse events.
  Participants will be monitored for adverse events during the study and for at least 30 days after the end of treatment.
  Analysis of toxicity following the completion of Stage 1, taking into consideration that Stage 2 will use lower doses of AZD5363, and at the end of Stage 2.

CONTACTS AND LOCATIONS:
Overall Officials: John FR Robertson, MD, Study Chair — University of Nottingham
Locations (11):
- United Kingdom (11):
  - Royal Derby Hospital, Derby, Derbyshire
  - Plymouth Hospitals NHS Trust, Derriford, Plymouth, Devon
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Poole Hospital NHS Foundation Trust, Poole, Dorset
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Western General Hospital, Edinburgh, Lothian
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - Kingsmill Hospital, Sutton in Ashfield, Nottinghamshire
  - Sheffield Cancer Research Centre, Sheffield, South Yorkshire
  - University Hospital Birmingahm, Birmingham, West Midlands
  - Leeds St James Institue of Oncology, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No